CLINICAL TRIAL: NCT04993664
Title: Influence of Pelacarsen on Arterial Wall Properties and Risk Factors in Patients After Myocardial Infarction With High Lp(a) Values
Brief Title: Influence of Pelacarsen on Patients After Myocardial Infarction With High Lp(a) Values (PEMILA)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative reason
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miran Sebestjen, Professor, principal investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEMILA
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Acute Coronary Syndrome; Lipoproteinemia; Inflammation; Genetic Polymorphisms
Keywords: Coronary heart disease; Acute coronary syndrome; Lipoprotein (a); Genetics; Secondary prevention; Endothelium; Inflammation; Genetic polymorphisms; NO synthetase; Dyslipidemia
MeSH Terms: conditions — Acute Coronary Syndrome; Inflammation; Coronary Disease; Dyslipidemias | interventions — pelacarsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelacarsen group (TQJ230) (Experimental): The first group will receive 80 mg of pelacarsen every month subcutaneously for 6 months.
  Interventions: Drug: Pelacarsen (TQJ230)
- Placebo group (Placebo Comparator): The first group will receive 80 mg of placebo every month subcutaneously for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pelacarsen (TQJ230) — The first group will receive pelacarsen. Blood samples from all patients will be drawn for laboratory measurements and genetics determination. Ultrasound measurement of endothelium-dependent dilatation of the brachial artery and beta stiffness of carotid arteries will be measured.
  Arms: Pelacarsen group (TQJ230)
Drug: Placebo — The second group will receive placebo. Blood samples from all patients will be drawn for laboratory measurements and genetics determination. Ultrasound measurement of endothelium-dependent dilatation of the brachial artery and beta stiffness of carotid arteries will be measured.
  Arms: Placebo group

SUMMARY:
The aim of study is to examine the relationship between lipid subfractions, inflammation and structural-functional properties of the arterial wall in patients after myocardial infarction with high lipoprotein (a) (Lp (a)) levels, to study genetic polymorphisms that determine lipid subfractions concentration on the functional and morphological properties of the arterial vascular wall in patients after myocardial infarction with high Lp (a) levels, to study the effect of pelacarsen on lipid subfractions, inflammation and structural-functional properties of arterial wall in patients after myocardial infarction with high Lp (a) levels and to study the influence of NOS-3 gene expression on the functional and morphological properties of the arterial vascular wall in the same patients.

Impaired blood fat metabolism and chronic inflammation represent possible causes of atherosclerosis. Lp (a) is an independent risk factor for cardiovascular disease and a prognostic predictor in patients after myocardial infarction. Despite recommended screening for elevated Lp (a), there is no specific drug treatment approved to reduce cardiovascular risk through lowering Lp (a). Besides subtilisin-kexin convertase type 9 (PCSK9) inhibitors, antisense oligonucleotides (ASOs) are currently only therapeutic agents that significantly reduce serum Lp (a) concentration. Pelacarsen by using an ASO directed against the messenger ribonucleic acid (mRNA) of apolipoprotein (a), reduces the production of apolipoprotein (a) in the liver and thus, the level of Lp (a).

However, there are no data on the relationship between Lp (a) values and polymorphisms for Lp (a), indicators of inflammation and impaired arterial function, and response to treatment with pelacarsen in patients after myocardial infarction with extremely high Lp (a) levels.

DETAILED DESCRIPTION:
Impaired blood fat metabolism and chronic inflammation represent possible causes of atherosclerosis. The early stage of the atherosclerosis process is characterized by endothelial cell damage, which results in impaired release and function of nitric oxide (NO) from the endothelium. NO is formed by endothelial NO synthetase (NOS-3) from the amino acid L-arginine, which is most pronounced in the vascular wall and is also most important in the process of atherosclerosis. The NOS-3 gene is located on chromosome 7; in the region 7q35-7q36. Functional polymorphisms are those that alter the expression or activity of NOS-3. Among functional polymorphisms, rs2070744, rs3918226 and rs1799983 single nucleotide polymorphisms (SNP) are important. Variations in the NOS-3 genes cause diversity in NO bioavailability and are responsible for endothelial dysfunction.

Lipoprotein (a) (Lp (a)) is a specific subfraction of lipoprotein that is an independent risk factor for cardiovascular disease and predicts the residual risk in patients with pre-existing atherosclerosis, regardless of serum LDL-cholesterol concentration. Circulating levels of Lp(a) are mainly genetically determined and varies according to ethnic group. Lp(a) has atherosclerotic, prothrombotic and pro-inflammatory effects. The gene encoding apo (a); LPA, is located on the long arm of chromosome 6 (6q2,6-2,7) and most variants in Lp (a) can be explained by genetic diversity in LPA. To date, the most studied genetic variant is the Kringle-IV type-2 (KIV2) polymorphism, which explains 30-70% of the diversity in Lp (a) in the population. Some KIV2 replicates are associated with smaller isoforms and higher plasma concentrations of Lp (a) which are causally and independently associated with coronary heart disease. Within LPA, the number of KIV2 copies, as well as one nucleotide polymorphism (SNP), rs3798220 and rs10455872, are associated with Lp (a) concentration and coronary heart disease. Besides subtilisin-kexin convertase type 9 (PCSK9) inhibitors, antisense oligonucleotides (ASOs) are currently only therapeutic agents that significantly reduce serum Lp (a) concentration and that have shown effectiveness in clinical trials, to provide reductions in cardiovascular morbidity and mortality. Pelacarsen by using an ASO directed against the mRNA of apolipoprotein (a), reduces the production of apolipoprotein (a) in the liver and thus, the level of Lp (a).

A 6-month randomized, double-blind, parallel group and placebo-controlled study will include 60 patients with established cardiovascular disease (CVD) (including myocardial infarction, ischemic stroke or symptomatic peripheral artery disease) and Lp (a) levels above 700 mg / L.

The investigators will do anamnesis, targeted clinical examination, take blood samples for laboratory measurements, ultrasound measure endothelium-dependent dilatation of the brachial artery and beta stiffness of carotid arteries. Patients will be divided into two groups according to the randomization list. The first group will receive pelacarsen 80 mg subcutaneously and the second group will receive corresponding placebo. After 6 months, the investigators will repeat all the mentioned investigations. Patients will be informed about the purpose and course of the study before starting the study. All patients will participate voluntarily, without pressure or inappropriate instigation and will give consent by signing the consent form.

The investigators hypotheses that in patients after myocardial infarction and high levels of Lp (a), Lp (a) and Lp (a) polymorphisms are associated with indicators of inflammation and structural-functional properties of the arterial wall; in patients after myocardial infarction and extremely high levels of Lp (a), pelacarsen reduces the value of Lp (a), indicators of inflammation and structural and functional involvement of the arterial wall; in patients after myocardial infarction and extremely high levels of Lp (a), the influence of pelacarsen on Lp (a), indicators of inflammation and structural-functional properties of the arterial wall depends on the presence of specific polymorphisms for Lp (a).

ELIGIBILITY:
Inclusion Criteria:

* concentration Lp (a) above 700 mg / L,
* optimally treated risk factors for cardiovascular events according to currently valid guidelines,
* history of myocardial infarction having occurred in the period 3 months to 10 years prior to the screening visit and / or
* history of ischemic stroke having occurred in the period 3 months to 10 years prior to the screening visit and / or
* clinically significant symptomatic peripheral artery disease.

Exclusion Criteria:

* uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and / or diastolic blood pressure ≥ 100 mmHg),
* heart failure New York Heart Association (NYHA) class IV,
* history of malignancy of any organ system,
* history of hemorrhagic stroke or other major bleeding,
* platelet count <140,000 per mm3,
* active liver disease or hepatic dysfunction (elevated transaminases above 3 times the norm, elevated bilirubin above 2 times the norm, elevated creatinine kinase above 3 times the norm),
* significant kidney disease (oGFR <30 ml / min),
* pregnant or nursing women,
* life expectancy less than 5 years,
* unwillingness to participate or lack of availability for follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasound functional and morphological properties of the arterial wall and Lp (a) concentration | Baseline
  Functional and morphological characteristics of arterial wall will correlate to Lp (a) concentrations.
Concentration of Lp (a) and SNP in the LPA gene | Baseline
  The serum concentration of Lp (a) will correlate with single nucleotide polymorphisms (SNP) in the LPA gene.
The effect of pelacarsen on functional and morphological properties of arterial wall after 6 months | Baseline
  Pelacarsen will improve functional and morphological properties of arterial wall. The investigators expect the improvements will be in correlation with the decrease of Lp (a) concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Miran Šebeštjen, prof., PhD, Study Chair — University Medical Centre Ljubljana (Slovenia); Sabina Ugovšek, MD, Principal Investigator — University Medical Centre Ljubljana (Slovenia)
Locations (1):
- University Medical Centre Ljubljana-Department of Vascular diseases and dept. of Cardiology, Ljubljana, Slovenia

REFERENCES:
- [Background] Pagidipati NJ, Gaziano TA. Estimating deaths from cardiovascular disease: a review of global methodologies of mortality measurement. Circulation. 2013 Feb 12;127(6):749-56. doi: 10.1161/CIRCULATIONAHA.112.128413. No abstract available. PMID 23401116
- [Background] McGill HC Jr, McMahan CA, Herderick EE, Malcom GT, Tracy RE, Strong JP. Origin of atherosclerosis in childhood and adolescence. Am J Clin Nutr. 2000 Nov;72(5 Suppl):1307S-1315S. doi: 10.1093/ajcn/72.5.1307s. PMID 11063473
- [Background] Wang JC, Bennett M. Aging and atherosclerosis: mechanisms, functional consequences, and potential therapeutics for cellular senescence. Circ Res. 2012 Jul 6;111(2):245-59. doi: 10.1161/CIRCRESAHA.111.261388. PMID 22773427
- [Background] Egashira K. Clinical importance of endothelial function in arteriosclerosis and ischemic heart disease. Circ J. 2002 Jun;66(6):529-33. doi: 10.1253/circj.66.529. PMID 12074266
- [Background] Bisoendial RJ, Kastelein JJ, Stroes ES. C-reactive protein and atherogenesis: from fatty streak to clinical event. Atherosclerosis. 2007 Dec;195(2):e10-8. doi: 10.1016/j.atherosclerosis.2007.04.053. Epub 2007 Jul 31. PMID 17669411
- [Background] Giles TD, Sander GE, Nossaman BD, Kadowitz PJ. Impaired vasodilation in the pathogenesis of hypertension: focus on nitric oxide, endothelial-derived hyperpolarizing factors, and prostaglandins. J Clin Hypertens (Greenwich). 2012 Apr;14(4):198-205. doi: 10.1111/j.1751-7176.2012.00606.x. PMID 22458740
- [Background] Tada H, Takamura M, Kawashiri MA. Lipoprotein(a) as an Old and New Causal Risk Factor of Atherosclerotic Cardiovascular Disease. J Atheroscler Thromb. 2019 Jul 1;26(7):583-591. doi: 10.5551/jat.RV17034. Epub 2019 Apr 30. PMID 31061262
- [Background] Machado-Silva W, Alfinito-Kreis R, Carvalho LS, Quinaglia-E-Silva JC, Almeida OL, Brito CJ, Ferreira AP, Cordova C, Sposito AC, Nobrega OT; Brasilia Heart Study Group. Endothelial nitric oxide synthase genotypes modulate peripheral vasodilatory properties after myocardial infarction. Gene. 2015 Sep 1;568(2):165-9. doi: 10.1016/j.gene.2015.05.042. Epub 2015 May 20. PMID 26002446
- [Background] Marsden PA, Heng HH, Scherer SW, Stewart RJ, Hall AV, Shi XM, Tsui LC, Schappert KT. Structure and chromosomal localization of the human constitutive endothelial nitric oxide synthase gene. J Biol Chem. 1993 Aug 15;268(23):17478-88. PMID 7688726
- [Background] Oliveira-Paula GH, Lacchini R, Tanus-Santos JE. Endothelial nitric oxide synthase: From biochemistry and gene structure to clinical implications of NOS3 polymorphisms. Gene. 2016 Jan 10;575(2 Pt 3):584-99. doi: 10.1016/j.gene.2015.09.061. Epub 2015 Sep 28. PMID 26428312
- [Background] Hingorani AD, Liang CF, Fatibene J, Lyon A, Monteith S, Parsons A, Haydock S, Hopper RV, Stephens NG, O'Shaughnessy KM, Brown MJ. A common variant of the endothelial nitric oxide synthase (Glu298-->Asp) is a major risk factor for coronary artery disease in the UK. Circulation. 1999 Oct 5;100(14):1515-20. doi: 10.1161/01.cir.100.14.1515. PMID 10510054
- [Background] Bostom AG, Cupples LA, Jenner JL, Ordovas JM, Seman LJ, Wilson PW, Schaefer EJ, Castelli WP. Elevated plasma lipoprotein(a) and coronary heart disease in men aged 55 years and younger. A prospective study. JAMA. 1996 Aug 21;276(7):544-8. doi: 10.1001/jama.1996.03540070040028. PMID 8709403
- [Background] Schaefer EJ, Lamon-Fava S, Jenner JL, McNamara JR, Ordovas JM, Davis CE, Abolafia JM, Lippel K, Levy RI. Lipoprotein(a) levels and risk of coronary heart disease in men. The lipid Research Clinics Coronary Primary Prevention Trial. JAMA. 1994 Apr 6;271(13):999-1003. doi: 10.1001/jama.1994.03510370051031. PMID 8139085
- [Background] Willeit P, Ridker PM, Nestel PJ, Simes J, Tonkin AM, Pedersen TR, Schwartz GG, Olsson AG, Colhoun HM, Kronenberg F, Drechsler C, Wanner C, Mora S, Lesogor A, Tsimikas S. Baseline and on-statin treatment lipoprotein(a) levels for prediction of cardiovascular events: individual patient-data meta-analysis of statin outcome trials. Lancet. 2018 Oct 13;392(10155):1311-1320. doi: 10.1016/S0140-6736(18)31652-0. Epub 2018 Oct 4. PMID 30293769
- [Background] Berthold HK, Gouni-Berthold I. Hyperlipoproteinemia(a): clinical significance and treatment options. Atheroscler Suppl. 2013 Jan;14(1):1-5. doi: 10.1016/j.atherosclerosissup.2012.10.037. PMID 23357133
- [Background] Hoover-Plow J, Huang M. Lipoprotein(a) metabolism: potential sites for therapeutic targets. Metabolism. 2013 Apr;62(4):479-91. doi: 10.1016/j.metabol.2012.07.024. Epub 2012 Oct 4. PMID 23040268
- [Background] Kamstrup PR, Tybjaerg-Hansen A, Steffensen R, Nordestgaard BG. Genetically elevated lipoprotein(a) and increased risk of myocardial infarction. JAMA. 2009 Jun 10;301(22):2331-9. doi: 10.1001/jama.2009.801. PMID 19509380
- [Background] Nordestgaard BG, Chapman MJ, Ray K, Boren J, Andreotti F, Watts GF, Ginsberg H, Amarenco P, Catapano A, Descamps OS, Fisher E, Kovanen PT, Kuivenhoven JA, Lesnik P, Masana L, Reiner Z, Taskinen MR, Tokgozoglu L, Tybjaerg-Hansen A; European Atherosclerosis Society Consensus Panel. Lipoprotein(a) as a cardiovascular risk factor: current status. Eur Heart J. 2010 Dec;31(23):2844-53. doi: 10.1093/eurheartj/ehq386. Epub 2010 Oct 21. PMID 20965889
- [Background] Lawn RM. How often has Lp(a) evolved? Clin Genet. 1996 Apr;49(4):167-74. doi: 10.1111/j.1399-0004.1996.tb03281.x. PMID 8828980
- [Background] Emerging Risk Factors Collaboration; Erqou S, Kaptoge S, Perry PL, Di Angelantonio E, Thompson A, White IR, Marcovina SM, Collins R, Thompson SG, Danesh J. Lipoprotein(a) concentration and the risk of coronary heart disease, stroke, and nonvascular mortality. JAMA. 2009 Jul 22;302(4):412-23. doi: 10.1001/jama.2009.1063. PMID 19622820
- [Background] Maranhao RC, Carvalho PO, Strunz CC, Pileggi F. Lipoprotein (a): structure, pathophysiology and clinical implications. Arq Bras Cardiol. 2014 Jul;103(1):76-84. doi: 10.5935/abc.20140101. PMID 25120086
- [Background] Ma L, Chan DC, Ooi EMM, Barrett PHR, Watts GF. Fractional turnover of apolipoprotein(a) and apolipoprotein B-100 within plasma lipoprotein(a) particles in statin-treated patients with elevated and normal Lp(a) concentration. Metabolism. 2019 Jul;96:8-11. doi: 10.1016/j.metabol.2019.04.010. Epub 2019 Apr 14. PMID 30995439
- [Background] Marcovina SM, Albers JJ. Lipoprotein (a) measurements for clinical application. J Lipid Res. 2016 Apr;57(4):526-37. doi: 10.1194/jlr.R061648. Epub 2015 Dec 4. PMID 26637278
- [Background] Tsimikas S. A Test in Context: Lipoprotein(a): Diagnosis, Prognosis, Controversies, and Emerging Therapies. J Am Coll Cardiol. 2017 Feb 14;69(6):692-711. doi: 10.1016/j.jacc.2016.11.042. PMID 28183512
- [Background] Rehberger Likozar A, Zavrtanik M, Sebestjen M. Lipoprotein(a) in atherosclerosis: from pathophysiology to clinical relevance and treatment options. Ann Med. 2020 Aug;52(5):162-177. doi: 10.1080/07853890.2020.1775287. Epub 2020 Jun 8. PMID 32453609
- [Background] Helgadottir A, Gretarsdottir S, Thorleifsson G, Holm H, Patel RS, Gudnason T, Jones GT, van Rij AM, Eapen DJ, Baas AF, Tregouet DA, Morange PE, Emmerich J, Lindblad B, Gottsater A, Kiemeny LA, Lindholt JS, Sakalihasan N, Ferrell RE, Carey DJ, Elmore JR, Tsao PS, Grarup N, Jorgensen T, Witte DR, Hansen T, Pedersen O, Pola R, Gaetani E, Magnadottir HB, Wijmenga C, Tromp G, Ronkainen A, Ruigrok YM, Blankensteijn JD, Mueller T, Wells PS, Corral J, Soria JM, Souto JC, Peden JF, Jalilzadeh S, Mayosi BM, Keavney B, Strawbridge RJ, Sabater-Lleal M, Gertow K, Baldassarre D, Nyyssonen K, Rauramaa R, Smit AJ, Mannarino E, Giral P, Tremoli E, de Faire U, Humphries SE, Hamsten A, Haraldsdottir V, Olafsson I, Magnusson MK, Samani NJ, Levey AI, Markus HS, Kostulas K, Dichgans M, Berger K, Kuhlenbaumer G, Ringelstein EB, Stoll M, Seedorf U, Rothwell PM, Powell JT, Kuivaniemi H, Onundarson PT, Valdimarsson E, Matthiasson SE, Gudbjartsson DF, Thorgeirsson G, Quyyumi AA, Watkins H, Farrall M, Thorsteinsdottir U, Stefansson K. Apolipoprotein(a) genetic sequence variants associated with systemic atherosclerosis and coronary atherosclerotic burden but not with venous thromboembolism. J Am Coll Cardiol. 2012 Aug 21;60(8):722-9. doi: 10.1016/j.jacc.2012.01.078. PMID 22898070
- [Background] Clarke R, Peden JF, Hopewell JC, Kyriakou T, Goel A, Heath SC, Parish S, Barlera S, Franzosi MG, Rust S, Bennett D, Silveira A, Malarstig A, Green FR, Lathrop M, Gigante B, Leander K, de Faire U, Seedorf U, Hamsten A, Collins R, Watkins H, Farrall M; PROCARDIS Consortium. Genetic variants associated with Lp(a) lipoprotein level and coronary disease. N Engl J Med. 2009 Dec 24;361(26):2518-28. doi: 10.1056/NEJMoa0902604. PMID 20032323
- [Background] Chasman DI, Shiffman D, Zee RY, Louie JZ, Luke MM, Rowland CM, Catanese JJ, Buring JE, Devlin JJ, Ridker PM. Polymorphism in the apolipoprotein(a) gene, plasma lipoprotein(a), cardiovascular disease, and low-dose aspirin therapy. Atherosclerosis. 2009 Apr;203(2):371-6. doi: 10.1016/j.atherosclerosis.2008.07.019. Epub 2008 Jul 26. PMID 18775538
- [Background] Ober C, Nord AS, Thompson EE, Pan L, Tan Z, Cusanovich D, Sun Y, Nicolae R, Edelstein C, Schneider DH, Billstrand C, Pfaffinger D, Phillips N, Anderson RL, Philips B, Rajagopalan R, Hatsukami TS, Rieder MJ, Heagerty PJ, Nickerson DA, Abney M, Marcovina S, Jarvik GP, Scanu AM, Nicolae DL. Genome-wide association study of plasma lipoprotein(a) levels identifies multiple genes on chromosome 6q. J Lipid Res. 2009 May;50(5):798-806. doi: 10.1194/jlr.M800515-JLR200. Epub 2009 Jan 5. PMID 19124843
- [Background] Hobbs HH, White AL. Lipoprotein(a): intrigues and insights. Curr Opin Lipidol. 1999 Jun;10(3):225-36. doi: 10.1097/00041433-199906000-00005. PMID 10431659
- [Background] Hajjar KA, Gavish D, Breslow JL, Nachman RL. Lipoprotein(a) modulation of endothelial cell surface fibrinolysis and its potential role in atherosclerosis. Nature. 1989 May 25;339(6222):303-5. doi: 10.1038/339303a0. PMID 2524666
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Anderson TJ, Gregoire J, Pearson GJ, Barry AR, Couture P, Dawes M, Francis GA, Genest J Jr, Grover S, Gupta M, Hegele RA, Lau DC, Leiter LA, Lonn E, Mancini GB, McPherson R, Ngui D, Poirier P, Sievenpiper JL, Stone JA, Thanassoulis G, Ward R. 2016 Canadian Cardiovascular Society Guidelines for the Management of Dyslipidemia for the Prevention of Cardiovascular Disease in the Adult. Can J Cardiol. 2016 Nov;32(11):1263-1282. doi: 10.1016/j.cjca.2016.07.510. Epub 2016 Jul 25. PMID 27712954
- [Background] O'Donoghue ML, Fazio S, Giugliano RP, Stroes ESG, Kanevsky E, Gouni-Berthold I, Im K, Lira Pineda A, Wasserman SM, Ceska R, Ezhov MV, Jukema JW, Jensen HK, Tokgozoglu SL, Mach F, Huber K, Sever PS, Keech AC, Pedersen TR, Sabatine MS. Lipoprotein(a), PCSK9 Inhibition, and Cardiovascular Risk. Circulation. 2019 Mar 19;139(12):1483-1492. doi: 10.1161/CIRCULATIONAHA.118.037184. PMID 30586750
- [Background] Tsimikas S, Moriarty PM, Stroes ES. Emerging RNA Therapeutics to Lower Blood Levels of Lp(a): JACC Focus Seminar 2/4. J Am Coll Cardiol. 2021 Mar 30;77(12):1576-1589. doi: 10.1016/j.jacc.2021.01.051. PMID 33766265
- [Background] Tsimikas S, Karwatowska-Prokopczuk E, Gouni-Berthold I, Tardif JC, Baum SJ, Steinhagen-Thiessen E, Shapiro MD, Stroes ES, Moriarty PM, Nordestgaard BG, Xia S, Guerriero J, Viney NJ, O'Dea L, Witztum JL; AKCEA-APO(a)-LRx Study Investigators. Lipoprotein(a) Reduction in Persons with Cardiovascular Disease. N Engl J Med. 2020 Jan 16;382(3):244-255. doi: 10.1056/NEJMoa1905239. Epub 2020 Jan 1. PMID 31893580